CLINICAL TRIAL: NCT02674750
Title: Open-Label, Phase 2 Study to Evaluate the Efficacy and Safety of CUDC-907 in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma, Including Patients With MYC Alterations
Brief Title: Study to Evaluate the Efficacy and Safety of CUDC-907 in Patients With RR DLBCL, Including Patients With MYC Alterations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Curis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUDC-907-201
Record Dates: First submitted 2016-01-29; First posted 2016-02-04 (Estimated); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Relapsed and/or Refractory Diffuse Large B-cell Lymphoma Including With Myc Alterations
Keywords: DLBCL; MYC
MeSH Terms: interventions — CUDC-907

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): Group A: MYC translocation+ and/or MYC gene copy number gain by FISH
  Interventions: Drug: CUDC-907
- Group B (Experimental): Group B: MYC expression in > 40% of tumor cells by IHC
  Interventions: Drug: CUDC-907
- Group C (Experimental): Group C: MYC translocation- by FISH, and MYC expression in < 40% of tumor cells, and no MYC gene copy number gain by FISH
  Interventions: Drug: CUDC-907

INTERVENTIONS:
Drug: CUDC-907

SUMMARY:
This is a Phase 2, open-label, multicenter trial designed to evaluate the efficacy and safety of CUDC-907 in subjects 18 years and older with Relapsed/Refractory (RR) MYC-altered Diffuse Large B-Cell Lymphoma (DLBCL).

DETAILED DESCRIPTION:
Patients with RR DLBCL will be eligible for treatment with CUDC-907, as long as they have tumor tissue available that can be tested for MYC-altered disease based on one of the following:

* Fresh tumor tissue obtained from biopsy accessible lesions , or
* Archived tumor tissue (most recent available)

Subjects will be required to submit archival tumor samples (most recent available) or fresh tumor samples for central FISH and IHC testing. Subjects whose tumors have been previously characterized as MYC-altered are strongly encouraged to enter the study. For subjects who enter the study with unconfirmed MYC-altered disease, fresh tumor samples are preferred.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. At least 2 but no more than 4 prior lines of therapy for the treatment of de novo DLBCL and ineligible for (or failed) autologous or allogeneic stem cell transplant (SCT) (salvage therapy, conditioning therapy and maintenance with transplant will be considered one prior treatment). NOTE: For follicular lymphoma transformed to DLBCL (t-FL/DLBCL), single agent non-cytotoxic therapy will not be considered as a line of therapy.
3. Histopathologically confirmed diagnosis of one of the following:

   * RR DLBCL per the 2008 World Health Organization (WHO) classification of hematopoietic and lymphoid tumors (Swerdlow et al, 2008).
   * High grade B-cell lymphoma (HGBL), with MYC and BCL2 and/or BCL6 rearrangements or DLBCL, NOS per the 2016 revision of the WHO classification of lymphoid neoplasms (Swerdlow et al, 2016).
   * Diagnosis of t-FL/DLBCL is allowed. However, other B-cell lymphomas including other transformed indolent lymphomas/DLBCL per the 2008 WHO classification, and Burkitt lymphoma are not eligible.

Exclusion Criteria:

1. Known primary mediastinal, ocular, epidural, testicular or breast DLBCL.
2. Active CNS involvement of their malignancy.
3. Known allergy or hypersensitivity to phosphatidylinositol 3 kinase (PI3K) inhibitors or any component of the formulations used in this study.
4. Cytotoxic anticancer therapy (e.g., alkylating agents, anti-metabolites, purine analogues) or any other systemic anticancer therapy within 2 weeks of study entry.
5. Radiotherapy delivered to non-target lesions within one week prior to starting study treatment or delivered to target lesions that will be followed on the study (note: prior sites of radiation will be recorded).
6. Treatment with experimental therapy within 5 terminal half-lives (t1/2) or 4 weeks prior to enrollment, whichever is longer.
7. Current or planned glucocorticoid therapy, with the following exceptions:

   * Doses ≤ 10 mg/kg/day prednisolone or equivalent is allowed, provided that the steroid dose has been stable or tapering for at least 14 days prior to the first dose of CUDC-907.
   * Inhaled, intranasal, intraarticular, and topical steroids are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-07; Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (20):
  - University of California San Francisco-Fresno, Fresno, California
  - University of Southern California, Norris Comprehensive Cancer Center, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Rochester, Rochester, New York
  - University of Oklahoma Health Sciences Center (OUHSC), Oklahoma City, Oklahoma
  - Cancer Care Associates, Tulsa, Oklahoma
  - Penn State Hershey Cancer Institute-Clinical Trials Office, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Tennessee Cancer Center, Knoxville, Tennessee
  - Tennessee Oncology Sarah Cannon, Nashville, Tennessee
  - Charles A. Sammons Cancer Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Durán i Reynals, Servicio de Oncología, Barcelona
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adverse Events were collected from signing of the ICF through the last patient visit. (July2016 - May 2019)
Groups:
- Group A: MYC translocation+ and/or MYC gene copy number gain by FISH
- Group B: MYC expression in > 40% of tumor cells by IHC
- Group C: MYC translocation- by FISH, and MYC expression in < 40% of tumor cells, and no MYC gene copy number gain by FISH
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 5 | 49 | 16
Completed (Completed = subjects stopped when Sponsor stopped study.) | 0 | 4 | 4
Not Completed | 5 | 45 | 12
Not completed — Death | 4 | 5 | 8
Not completed — Lost to Follow-up | 0 | 8 | 0
Not completed — Lack of Efficacy | 1 | 17 | 3
Not completed — Withdrawal by Subject | 0 | 7 | 1
Not completed — Other | 0 | 8 | 0

BASELINE CHARACTERISTICS:
Population: ITT (Intent to Treat)
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 5 | 49 | 16 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 29 | 8 | 40
  >=65 years | 2 | 20 | 8 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 20 | 7 | 29
  Male | 3 | 29 | 9 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 1 | 6
  Not Hispanic or Latino | 3 | 44 | 14 | 61
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 3
  White | 4 | 44 | 14 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 4 | 42 | 15 | 61
  Spain | 0 | 2 | 1 | 3
  France | 1 | 5 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Efficacy of CUDC-907 in subjects with Relapsed/Refractory MYC-altered Diffuse Large B-Cell Lymphoma (DLBCL)
Time Frame: 2 Years
Population: The analysis of ORR was not performed since central radiographic review was not performed, due to inconclusive efficacy at the interim analysis, enrollment was permanently stopped in August 2017.
Groups:
- CUDC-907: RR-DLBCL, including with MYC alterations detected by FISH or by >=40% MYC by IHC
  CUDC-907
Arm/Group | CUDC-907
Number analyzed (Participants) | 0

2. Secondary Outcome: Median Progression-free Survival
Description: Efficacy of CUDC-907 in subjects with Relapsed/Refractory MYC-altered DLBCL
Time Frame: 1 year
Population: Evaluable population; The number of participants in this table include the evaluable participants which is different from the overall number of participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 2 | 28 | 9
months | 1.2 [1.02 to 1.41] | 2.7 [1.28 to 4.05] | 2.6 [1.28 to 21.94]

3. Secondary Outcome: Overall Survival (OS)
Description: Efficacy of CUDC-907 in subjects with Relapsed/Refractory MYC-altered DLBCL
Time Frame: 1 year
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 2 | 28 | 9
participants | 1 | 17 | 2

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Efficacy of CUDC-907 in subjects with Relapsed/Refractory MYC-altered DLBCL Note: Response is defined using Cheson 2007 criteria. CR=Complete Response; PR=Partial Response; SD=Stable Disease. a. Two-sided exact binomial 95% confidence interval. Revised Response Criteria for Malignant Lymphoma (Cheson 2007) was used for the assessment of response. DCR is defined as the proportion of patients having best response of complete response, partial response, or stable disease.
Time Frame: 1 year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 2 | 28 | 9
percentage of participants | 0.0 [0.00 to 84.19] | 46.4 [27.51 to 66.13] | 44.4 [13.70 to 78.80]

5. Secondary Outcome: Number of Participants and Severity of Adverse Events (AEs), Serious Adverse Events (SAEs), and Other Safety Parameters
Description: Number of participants and severity of adverse events (AEs), serious adverse events (SAEs), and other safety parameters in patients receiving CUDC-907.
Time Frame: AEs were collected for each participant for the duration that they remained on the study, on average of 4 months
Population: Safety Population; The number of participants in this table include the participants evaluable for safety which is different from the overall number of participants.
Measure: Number; unit: participants
Arm/Group | CUDC-907
Number analyzed (Participants) | 68
participants
  Experienced at least 1 TEAE | 68
  Experienced at least 1 study tx-related TEAE | 59
  Experienced a Grade <3 TEAE | 52
  Experienced a Grade <3 TEAE tx-related | 34
  Experienced at least 1 tx emergent SAE | 30
  Experienced a TEAE with outcome of death | 17
  Experienced a TEAE leading to D/C | 11

ADVERSE EVENTS:
Time Frame: AEs were collected for each participant for the duration that they remained on the study, on average of 4 months
Arm/Group | CUDC-907
All-Cause Mortality (participants affected / at risk) | 17/68
Serious Adverse Events (participants affected / at risk) | 30/68
Other Adverse Events (participants affected / at risk) | 68/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CUDC-907 (N=68)
Acute Kidney Injury (Renal and urinary disorders) | 3 (3)
Asthenia (General disorders) | 1 (1)
Disease Progression (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Diffuse Large B Cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Diarhhea (Gastrointestinal disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Citrobacter Batremia (Infections and infestations) | 1 (1)
Cytomegalovirus (Infections and infestations) | 1 (1)
Enterococcal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
hyperbilirubenemia (Hepatobiliary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Gullain-Barre Syndrome (Nervous system disorders) | 1 (1)
Device occulsion (Product Issues) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CUDC-907 (N=68)
Diarrhea (Gastrointestinal disorders) | 49 (49)
Nausea (Gastrointestinal disorders) | 33 (33)
Vomiting (Gastrointestinal disorders) | 19 (19)
Constipation (Gastrointestinal disorders) | 14 (14)
Abdominal Pain (Gastrointestinal disorders) | 12 (12)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 24 (24)
Pyrexia (General disorders) | 13 (13)
Peripheral edema (General disorders) | 8 (8)
Asthensia (General disorders) | 5 (5)
Chills (General disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 37 (37)
Decreased appetite (Metabolism and nutrition disorders) | 23 (23)
Hypomagnesia (Metabolism and nutrition disorders) | 27 (27)
Dehydration (Metabolism and nutrition disorders) | 19 (19)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (12)
Hyperuricemia (Metabolism and nutrition disorders) | 13 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 28 (28)
Anemia (Blood and lymphatic system disorders) | 18 (18)
Neutropenia (Blood and lymphatic system disorders) | 14 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Dizziness (Nervous system disorders) | 13 (13)
Headache (Nervous system disorders) | 6 (6)
Dysgeusia (Nervous system disorders) | 5 (5)
Upper Respiratory Infection (Infections and infestations) | 6 (6)
Sepsis (Infections and infestations) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Acute Kidney Injury (Renal and urinary disorders) | 11 (11)
Diffuse Large B Cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
Due to inconclusive efficacy at the interim analysis, enrollment was permanently stopped in August 2017.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT02674750/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT02674750/ICF_001.pdf